CLINICAL TRIAL: NCT00003186
Title: Dynamic In Vivo Lymphography and Sentinel Node Biopsy in Colorectal Cancer: A Feasibility Study
Brief Title: Diagnostic Procedure for Identifying Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: DS 96-57; RPCI-DS-96-57; NCI-G98-1371
Record Dates: First submitted 1999-11-01; First posted 2004-05-19 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; adenocarcinoma of the colon; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — iso-sulfan blue; Sentinel Lymph Node Biopsy

INTERVENTIONS:
Drug: isosulfan blue
Procedure: lymphangiography
Procedure: sentinel lymph node biopsy

SUMMARY:
RATIONALE: Diagnostic procedures, such as lymphography, may improve the identification of patients with metastatic colorectal cancer.

PURPOSE: Clinical trial to study the effectiveness of lymphography in determining the presence or absence of metastatic colorectal cancer in patients.

DETAILED DESCRIPTION:
OBJECTIVES: I. Confirm that injection of isosulfan blue into the mucosa or serosa immediately adjacent to a colorectal cancer results in the lymphatic transport of that agent initially to a specific regional lymph node that can readily be identified on visual inspection, dissected, and histologically evaluated for the presence or absence of metastatic disease.

OUTLINE: All patients receive an injection of isosulfan blue into peritumor serosa upon intraoperative identification of the primary tumor, prior to mesenteric mobilization. If colonoscopy is otherwise indicated, the injection may be delivered to the peritumor mucosa via colonoscopy during the case. The mesentery adjacent to the injection is inspected and the lymphatic pattern and nodes demonstrated by the isosulfan blue are diagrammed and photographed. The sentinel node(s) are surgically dissected and evaluated. If needed, a second injection of isosulfan blue may be given. Prior to mobilization of liver for resection of metastases, isosulfan blue is injected subcapsularly around the metastatic lesion.

PROJECTED ACCRUAL: There will be 10 patients accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Patients must be undergoing surgical resection of a colorectal primary adenocarcinoma Metastatic colorectal cancer to liver (hepatic metastases) allowed

PATIENT CHARACTERISTICS: Age: 18 to 75 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No known or suspected allergy to isosulfan blue Not pregnant

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-04; Primary Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A. Rodriguez-Bigas, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Result] Kane JM 3rd, Kahlenberg MS, Rodriguez-Bigas MA, Gibbs JF, Petrelli NJ. Intraoperative hepatic lymphatic mapping in patients with liver metastases from colorectal carcinoma. Am Surg. 2002 Sep;68(9):745-50. PMID 12356141